CLINICAL TRIAL: NCT00548197
Title: Preoperative Injection of Bevacizumab Prior to Vitreoretinal Surgery in Diabetic Tractional Retinal Detachment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 85-A-57
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2007-02

CONDITIONS: Intravitreal Bevacizumab Injection; Pars Plana Vitrectomy; Tractional Retinal Detachment; Diabetic Retinopathy
Keywords: Intravitreal Bevacizumab injection; Pars plana vitrectomy; tractional retinal detachment; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intravitreal Bevacizumab will be injected 2.5 mg IVB 3-5 days before operation in diabetic patients who were candidates for vitrectomy before performing pars plana vitrectomy
  Interventions: Drug: Bevacizumab
- Control group (No Intervention): no injection before performing pars plana vitrectomy in diabetic patients who were candidates for vitrectomy

INTERVENTIONS:
Drug: Bevacizumab — one intravitreal injection of 2.5 mg Bevacizumab 3-5 days before performing pars plana vitrectomy
  Other Names: Brand name of Bevacizumab is Avastin
  Arms: Intervention group

SUMMARY:
Vitreoretinal surgery for epiretinal proliferation tractional retinal detachment associated with proliferative diabetic retinopathy (PDR) is often complicated by hemorrhage from fibrovascular tissue. To control the bleeding during tissue dissection multiple measures and techniques are used.

Bevacizumab is an anti VEGF antibody which has been used to induce regression of ocular neovascularization. Its intraocular injection has been increasingly used for treatment of choroidal neovascularization (CNV) associated with age related macular degeneration (AMD) with fairly good success.Also it has been shown to be effective for treatment of PDR complicated with vitreous hemorrhage and iris neovascularization. We hypothesized that if anti-angiogenic agents, such as bevacizumab are injected into the vitreous cavity before vitrectomy in cases of PDR; there may be partial regression of neovascularization resulting in less intraoperative (and postoperative) hemorrhage. This can make the operation easier and shorter and lessen the need for intraocular cautery..

In this study diabetic patients who are candidated for vitrectomy with similar complexity scores will be randomized to preoperative injection or no injection of 2.5 mg Bevacizumab .In the injection group, 2.5 mg of bevacizumab (0.1 ml of commercially available Avastin vial, Genentech, inc. South San Francisco, CA) will be injected into the vitreous 3-5 days before operation.

During each operation, the number of endodiathermy applications, backflush needle applications and the duration of surgery will be recorded by an independent observer. Also, type of tamponade, post operation vitreous hemorrhage and 3 months postoperative visual acuities wil be recorded. all these parameters will be compared in two groups.

DETAILED DESCRIPTION:
Eligibility criteria:

Diabetic tractional retinal detachment-complexity score between 4 and 8

Main outcome measures:

best corrected visual acuity-anatomic condition of the retine(re-attachment of the retina)

ELIGIBILITY:
Inclusion Criteria:

* Those patients with tractional retinal detachment who are candidated for pars plana vitrectomy.
* Complexity score between 4 and 8.

Exclusion Criteria:

* Previous vitreoretinal surgery.
* Presence of any other vitreoretinal pathology such as past or present uveitis, and retinal artery or vein occlusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Modarres, MD, Study Director — Iran University of Medical Sciences(IUMS)
Locations (1):
- Rasool Akram Hospital, Tehran, Iran

REFERENCES:
- [Background] Spaide RF, Fisher YL. Intravitreal bevacizumab (Avastin) treatment of proliferative diabetic retinopathy complicated by vitreous hemorrhage. Retina. 2006 Mar;26(3):275-8. doi: 10.1097/00006982-200603000-00004. PMID 16508426
- [Background] Castellarin A, Grigorian R, Bhagat N, Del Priore L, Zarbin MA. Vitrectomy with silicone oil infusion in severe diabetic retinopathy. Br J Ophthalmol. 2003 Mar;87(3):318-21. doi: 10.1136/bjo.87.3.318. PMID 12598446
- [Background] Grisanti S, Biester S, Peters S, Tatar O, Ziemssen F, Bartz-Schmidt KU; Tuebingen Bevacizumab Study Group. Intracameral bevacizumab for iris rubeosis. Am J Ophthalmol. 2006 Jul;142(1):158-60. doi: 10.1016/j.ajo.2006.02.045. PMID 16815268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Intravitreal Bevacizumab will be injected 2.5 mg IVB 3-5 days before operation in diabetic patients who were candidates for vitrectomy before performing pars plana vitrectomy
  Bevacizumab: one intravitreal injection of 2.5 mg Bevacizumab 3-5 days before performing pars plana vitrectomy
- Control: no injection before performing pars plana vitrectomy in diabetic patients who were candidates for vitrectomy
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.3) | 53.2 (11.7) | 54.63 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity
Description: Post operative best corrected visual acuity ( best distance vision with eyeglasses or contact lenses)
Time Frame: last follow up, an average of 7 months post-operation
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22 | 18
LogMar | 1.1 (0.4) | 1.4 (0.3)

2. Secondary Outcome: Anatomic Status of the Retina
Description: Number of Participants with Postoperative Vitreous Hemorrhage
Time Frame: Last follow up, an average of 7 months post-operation
Population: Postoperative Vitreous Hemorrhage
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 22 | 18
Participants | 0 | 7

ADVERSE EVENTS:
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=22) | Control (N=18)
Inferior rhegmatogenous retinal detachment and perisillicone proliferations (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No